CLINICAL TRIAL: NCT01983020
Title: Randomized Double Blind Comparison of Peri-Operative Standard Analgesia With Peri-Operative Lidocane, Ketamine, or Lidocane and Ketamine Combination, Infusion for Patients Undergoing Spine Surgery
Brief Title: Peri-Operative Lidocane, Ketamine, or Lidocane and Ketamine Combination, Infusion for Patients Undergoing Spine Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 073-10
Record Dates: First submitted 2013-11-07; First posted 2013-11-13 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ketamine (Experimental): Ketamine infused at 0.25 mg/kg/hour.
  Interventions: Drug: Ketamine
- Lidocaine (Experimental): Lidocaine infused at 0.5 mg/kg/hour.
  Interventions: Drug: Lidocaine
- Ketamine and Lidocaine (Experimental): Ketamine infused at 0.25 mg/kg/hour along with lidocaine at 0.5 mg/kg/hour
  Interventions: Drug: Lidocaine; Drug: Ketamine
- Placebo (Placebo Comparator): Placebo (saline) given to compare usual treatment against active agents in post operative pain management.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Lidocaine
  Arms: Ketamine and Lidocaine; Lidocaine
Drug: Ketamine
  Arms: Ketamine; Ketamine and Lidocaine
Other: Saline
  Arms: Placebo

SUMMARY:
This study has been designed as a controlled clinical trial to evaluate the efficacy of brief lidocaine infusion, brief ketamine infusion and a lidocaine/ketamine combined infusion when added to conventional opioid therapy following major spine surgery, as well as to evaluate the effects of the lidocaine/ketamine pain protocol on the feasibility of performing routine intraoperative neurophysiology during spine surgery in adults and determine whether this infusion protocol is compatible with intraoperative neurophysiology on spine surgery patients. If one or more of the approaches is confirmed as efficacious and safe, it could have a significant impact on the routine management of postoperative pain in this context.

ELIGIBILITY:
Inclusion Criteria:

Male and Female >/= 18 years of age Patients undergoing first-time fusion surgery or surgery to revise a prior fusion Able to read, write and speak in English, and able to give informed consent for the study

Exclusion Criteria:

Any disease associated with major organ dysfunction renal dysfunction hepatic dysfunction cardiac dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Kaplan, MD, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Beth Israel Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine: Ketamine infused at 0.25 mg/kg/hour.
  Ketamine
- Lidocaine: Lidocaine infused at 0.5 mg/kg/hour.
  Lidocaine
- Ketamine and Lidocaine: Ketamine infused at 0.25 mg/kg/hour along with lidocaine at 0.5 mg/kg/hour
  Lidocaine
  Ketamine
Period: Overall Study
Arm/Group | Ketamine | Lidocaine | Ketamine and Lidocaine | Placebo
Started | 12 | 11 | 12 | 11
Completed | 12 | 11 | 12 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Lidocaine | Ketamine and Lidocaine | Placebo | Total
Number analyzed (Participants) | 12 | 11 | 12 | 11 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (11.85) | 55.16 (16.23) | 50.3 (11.5) | 56.3 (12.7) | 54.39 (13.08)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 12 | 11 | 46
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 8 | 8 | 31
  Male | 4 | 4 | 4 | 3 | 15
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 12 | 11 | 46

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity
Description: The primary outcome will be average pain intensity at rest on postoperative day 1 - 3. Pain Intensity rated from 0 (none) to 10 (severe).
Time Frame: postoperative day 1 - 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Lidocaine | Ketamine and Lidocaine | Placebo
Number analyzed (Participants) | 12 | 11 | 12 | 11
units on a scale | 6.29 (2.42) | 5.76 (2.25) | 5.51 (2.60) | 6.40 (2.59)

ADVERSE EVENTS:
Arm/Group | Ketamine | Lidocaine | Ketamine and Lidocaine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/11 | 3/12 | 1/11
Other Adverse Events (participants affected / at risk) | 2/12 | 2/11 | 6/12 | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=12) | Lidocaine (N=11) | Ketamine and Lidocaine (N=12) | Placebo (N=11)
Diplopia (Eye disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (8) | 1 (1)
Low Blood Pressure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=12) | Lidocaine (N=11) | Ketamine and Lidocaine (N=12) | Placebo (N=11)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cold Sweats (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Sedation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lightheadedness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Itching (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No